CLINICAL TRIAL: NCT02275871
Title: Dual-energy Contrast-enhanced Digital Subtraction Mammography (CESM) as a Tool to Screen High Risk Women for Breast Cancer: a Comparison to Screening Breast MRI
Brief Title: Comparison of Contrast-enhanced Spectral Mammography (CESM) to MRI in Screening High Risk Women for Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Didn't have funding to support the study design
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Jordana Phillips, MD, Principal Investigator, Beth Israel Deaconess Medical Center
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-225
Record Dates: First submitted 2014-10-20; First posted 2014-10-27 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRI and CESM (Experimental): High risk patients will get standard of care screening MRI and study CESM on the same day.
  Interventions: Other: MRI; Other: CESM

INTERVENTIONS:
Other: MRI — High risk screening MRI will be performed as part of the patient's routine care.
Other: CESM — After the MRI is complete, the patient will be brought to the mammography department for the contrast enhanced mammogram. The contrast enhanced mammogram will be independently interpreted by two study radiologists (randomly assigned) who are blinded to the MRI. They will then compare to the MRI to determine clinical follow-up. Any finding seen on MRI will be followed according to the MR protocol. Any finding seen on CESM only, will have a diagnostic work-up with mammography and ultrasound. If this work-up is negative, then follow-up CESM exams will be performed. Each patient will be followed for 2 years to determine sensitivity and specificity for both modalities.
  Other Names: Contrast Enhanced Spectral Mammography

SUMMARY:
This research study is comparing Dual-Energy Contrast-Enhanced Spectral Mammography (CESM) to MRI as a screening tool for breast cancer.

DETAILED DESCRIPTION:
This research study is being done to test how well a contrast enhanced mammogram compares to MRI in screening for breast cancer in people who are at higher risk for developing breast cancer.

Standard screening mammograms can miss breast cancers due to its inability to "see through" dense breast tissue. For this reason, women at increased risk for the development of breast cancer often undergo additional screening beyond conventional mammography with magnetic resonance imaging (MRI). Although screening MRI is very sensitive for finding breast cancer, it also finds many areas that are benign (not cancer). The only way to know which is the cancer is to perform a biopsy, which contributes to patient anxiety and leads to many unnecessary biopsies.

In the preliminary studies performed in women already diagnosed with breast cancer, contrast enhanced mammography was shown to have a similar sensitivity for finding primary breast cancer but detected fewer of the benign findings which would result in fewer unnecessary biopsies. It is also a faster and less expensive exam compared to MRI. Contrast mammography was FDA approved in 2011 and is used now as a tool to help work-up abnormalities seen on standard mammography and ultrasound.

We are now studying to see if contrast enhanced mammography will also be a beneficial tool in the screening setting to screen high risk patients for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age > or equal to 30 years
* High risk (>20% lifetime risk)
* Has a bilateral mammogram within the last 7 months
* Has had a same day high risk screening MRI

Exclusion Criteria:

* Participants who have a known allergy or contraindication to iodinated contrast.
* Participants who have a known allergy to food or medications.
* Participants who have renal insufficiency or failure.
* Participants who are pregnant or breastfeeding.
* Participants with a concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-11; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Number of cancers and false positive findings identified on CESM versus MRI as a measure of sensitivity and specificity | 4 years
  All CESM and MRI cases will be evaluated for the presence or absence of malignancy and will be coded to reflect this interpretation. Breast imaging-reporting and data system (BIRADS) scores of 1-3 represent the absence of malignancy and BIRADS code of 4-5 represent the presence of malignancy. These cases will be compared to the truth of whether malignancy developed in the patient based on biopsy results and long term clinical follow-up (2 years).

CONTACTS AND LOCATIONS:
Overall Officials: Jordana Phillips, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States